CLINICAL TRIAL: NCT00162747
Title: Topical Emollient Therapy for Prevention of Infections in Preterm Infants
Brief Title: Topical Therapy for Prevention of Infections in Preterm Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 98-04-21-03-2; H990772; 914-2123
Record Dates: First submitted 2005-09-07; First posted 2005-09-13 (Estimated); Last update posted 2005-09-13 (Estimated); Status verified 2005-06

CONDITIONS: Skin Diseases
Keywords: Pre-term infants; skin infections; infant skin; Aquaphor; sunflower seed oil; nutrition; skin care
MeSH Terms: conditions — Skin Diseases; Cellulitis | interventions — Petrolatum; Sunflower Oil

INTERVENTIONS:
Drug: Aquaphor
Drug: Sunflower Seed Oil

SUMMARY:
The purpose of this study is to determine how to best take care of the skin of preterm infants in order to prevent infections through the skin.

DETAILED DESCRIPTION:
The skin of babies who are born too early is not mature, which means they are at risk for infections of the skin or in the body. Their skin also become very dry, leading to cracking and breakdown, and this may feel painful or uncomfortable for the infant.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants

Exclusion Criteria:

* Full-term infant

Ages: 7 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600
Dates: Start 2001-12; Study Completion 2005-06

PRIMARY OUTCOMES:
Three weeks after application of the intervention, blood will be drawn from those enrolled in the control group.

SECONDARY OUTCOMES:
Atleast four additional times over the first four weeks of the child's life, the skin will be studied by lightly rubbing the skin with a cotton swab to detect germs on the skin and observing and recording the condition of the baby's skin.

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Darmstadt, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Dhaka Shishu Hospital, Dhaka, Bangladesh

REFERENCES:
- [Derived] Darmstadt GL, Khan NZ, Rosenstock S, Muslima H, Parveen M, Mahmood W, Ahmed ASMNU, Chowdhury MAKA, Zeger S, Saha SK. Impact of emollient therapy for preterm infants in the neonatal period on child neurodevelopment in Bangladesh: an observational cohort study. J Health Popul Nutr. 2021 May 26;40(1):24. doi: 10.1186/s41043-021-00248-9. PMID 34039435